CLINICAL TRIAL: NCT00029211
Title: A Randomized Controlled Trial of Echinacea in Children
Brief Title: A Trial of Echinacea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000114-01 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Echinacea extract

INTERVENTIONS:
Drug: Echinacea

SUMMARY:
This is a randomized trial to determine if echinacea is effective in shortening the length and/or lessening the severity of colds in children 2 through 11 years old.

DETAILED DESCRIPTION:
Upper respiratory tract infections (URI's) are a significant health burden in childhood. URI's are a major reason for visits to health care providers, and up to 35 percent of young children at any given time are taking some over-the-counter cold medication. Unfortunately, data suggest that most of these medications have limited effectiveness. Alternative medical therapies are growing in popularity; in a recent survey of parents of children being seen by pediatricians in Seattle, Washington, 24.2 percent indicated that their child had been seen by an alternative medicine health care provider, and 53.3 percent received therapies for the treatment of URI's in children. The proposed study is a randomized, double blind, placebo controlled trial of Echinacea for the treatment of URI's in children 2-11 years old. The aims of the project are: to determine if Echinacea shortens the duration and/or lessens the severity of URI's, if children receiving Echinacea for treatment of URI's have a reduced rate of secondary bacterial infections, and to determine if the use of Echinacea in patients 2-11 years old is associated with any significant side effects. A two-year study of 600 children is planned. Not only will the results of this study determine if Echinacea, the most popular medicinal herb sold in the United States, is an effective therapy for URI's in children, the study will provide a design framework for further assessment on the efficacy of other complementary and alternative medicines in children.

ELIGIBILITY:
Inclusion Criteria:

* Parent available to observe child during the night
* Parent peaks and reads English

Exclusion Criteria:

* History of asthma or allergic rhinitis
* History of auto-immune disease
* History of chronic lung disease
* Allergy to sunflower species

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600
Dates: Start 2000-04; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: James Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- Child Health Institute, University of Washington, Seattle, Washington, United States